CLINICAL TRIAL: NCT00094172
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of Atorvastatin in Patients With Clinically Isolated Syndrome and High Risk of Conversion to Multiple Sclerosis (ITN020AI)
Brief Title: Atorvastatin (Lipitor) Therapy in Patients With Clinically Isolated Syndrome (CIS) at Risk for Multiple Sclerosis
Acronym: STAYCIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAIT ITN020AI
Record Dates: First submitted 2004-10-14; First posted 2004-10-15 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: Early Multiple Sclerosis; MS; Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): 80 mg/day
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin at the dose of 80 mg/day. Participants will be allowed to decrease the daily dose to 40 mg/day if the higher dose is not well-tolerated
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo — tablet form
  Other Names: Placebo Treatment
  Arms: Placebo

SUMMARY:
Patients who have been diagnosed with clinically isolated syndrome (CIS) often develop problems related to the central nervous system, which controls the nerves in the body. Some of these patients may later be diagnosed with multiple sclerosis (MS), a progressive disease of the nervous system. The purpose of this study is to determine if the drug atorvastatin is helpful to CIS patients.

Study hypothesis: Early intervention with atorvastatin in patients with CIS will result in a state of immunological tolerance.

DETAILED DESCRIPTION:
CIS is a single clinical event indicating temporary disruption of normal nerve function. CIS patients may have a loss of vision in one eye; trouble with balance; double vision; numbness in the face; and tingling, numbness, or weakness in the arms or legs. Some CIS patients may develop MS, but others may not. Studies have shown that when CIS is accompanied by magnetic resonance imaging (MRI)-detected brain lesions that are consistent with those seen in MS, there is a high risk of a second neurologic event and a diagnosis of MS within several years. This study will evaluate the efficacy of atorvastatin, an antihyperlipidemic, in the prevention of MS in CIS patients.

This study will last 18 months. All participants must complete a 3- to 5-day course of corticosteroids at least 28 days before the baseline evaluations. This corticosteroid therapy must be initiated within 60 days of CIS onset. Participants will be randomly assigned to receive 80 mg of either atorvastatin or placebo by mouth daily for 12 months. Study visits will occur at screening and every 3 months thereafter until the end of the 18-month study. Blood collection will occur at selected visits, and other additional evaluations will be performed at Months 1 and 2. Selected participants will undergo MRI brain scans. Participants will be offered interferon beta-1a (Avonex®), free of charge, if they develop disease activity. Participants will be instructed to report any change in their health status to their treating physician within 48 hours of the onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinically isolated syndrome (CIS) as defined by an acute or subacute well-defined neurological event lasting at least 48 hours and consistent with MS (i.e., optic neuritis, spinal cord syndrome, brainstem/cerebellar syndromes). Other causes for optic neuritis other than CIS must be ruled out by an ophthalmologist. Patients with other "clinically silent" abnormal findings found upon neurological examination that are not attributable to the presenting symptom are not excluded.
* Onset of CIS symptoms occurring within 90 days of randomization
* Abnormal, unenhanced brain MRI with 2 or more clinically silent T2 lesions greater than or equal to 3 mm in diameter, at least one of which is periventricular in location or ovoid in shape
* Willing to use acceptable methods of contraception
* Have received 3 to 5 days of corticosteroid therapy within 60 days of CIS onset

Exclusion Criteria:

* Definite diagnosis of MS according to McDonald criteria
* Previous history of neurological symptoms lasting more than 48 hours. Patients with a history of neurological symptoms lasting less than 48 hours will not be excluded.
* Prior use of interferon, glatiramer acetate, cyclophosphamide, mitoxantrone, or plasmapheresis anytime prior to study entry
* Use of interferon preparations (unless as specified by the protocol), glatiramer acetate, cyclophosphamide, mitoxantrone, or plasmapheresis during the study
* Use of cyclosporine, fibric acid derivatives, niacin, erythromycin, or azole antifungal during the study
* Received more than 5 g of methylprednisolone (or the equivalent of other IV corticosteroid) prior to study screening
* Use of a cholesterol-lowering agent during the 3 months prior to study screening or need for such agents during the study
* Previous history of severe side effects with statin therapy
* Prior exposure to total lymphoid irradiation
* History of substance abuse in the 12 months prior to study screening
* History of systemic illness or medical condition that would limit the likelihood of completing the MRI procedures or would interfere with the measurement of a therapeutic effect
* Implanted pacemakers, cochlear implants, defibrillators, or metallic objects on or inside the body
* Uncontrolled hypertension, asthma, known malignancy other than skin cancer, symptomatic cardiac disease, epilepsy, insulin-dependent diabetes, or symptoms that can only be explained by systemic lupus erythematosus (SLE) or other autoimmune diseases
* Active liver disease
* Major medical illnesses or psychiatric impairment that in the investigator's opinion could interfere with the study
* History of severe depression or suicidal ideation within 1 year of study entry
* Pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Zamvil, MD, PhD, Study Chair — University of California, San Francisco; Emmanuelle Waubant, MD, PhD, Study Chair — University of California, San Francisco
Locations (14):
- United States (13):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Keck School of Medicine, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale MS Research Center, New Haven, Connecticut
  - Johns Hopkins, Baltimore, Maryland
  - Washington University Multiple Sclerosis Center, St Louis, Missouri
  - Jacobs Neurological Institute, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Mason MS Center, Seattle, Washington
- Montreal Neurological Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials available to the public.

REFERENCES:
- [Result] Waubant E, Pelletier D, Mass M, Cohen JA, Kita M, Cross A, Bar-Or A, Vollmer T, Racke M, Stuve O, Schwid S, Goodman A, Kachuck N, Preiningerova J, Weinstock-Guttman B, Calabresi PA, Miller A, Mokhtarani M, Ikle D, Murphy S, Kopetskie H, Ding L, Rosenberg E, Spencer C, Zamvil SS; ITN STAyCIS Study Group; ITN020AI Study Management Team. Randomized controlled trial of atorvastatin in clinically isolated syndrome: the STAyCIS study. Neurology. 2012 Apr 10;78(15):1171-8. doi: 10.1212/WNL.0b013e31824f7fdd. Epub 2012 Mar 28. PMID 22459680
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY547 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY547 — ImmPort study identifier is SDY547. ImmPort is the long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
- Available data/document: Study summary, -design with synopsis, -adverse events, -medications, -demographics, -lab tests, -files et al.: SDY547 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY547 — ImmPort study identifier is SDY547
- Available data/document: Individual Participant Data Set: ITN020AI — http://www.itntrialshare.org/project/Studies/ITN020AIPUBLIC/Study%20Data/begin.view? — TrialShare study identifier is ITN020AI
- Available data/document: Study overview with synopsis, -navigator, -schedule of assessments, data and reports, -manuscripts and abstracts et al.: ITN020AI — http://www.itntrialshare.org/project/Studies/ITN020AIPUBLIC/Study%20Data/begin.view? — TrialShare is the research portal of the Immune Tolerance Network (ITN) that makes data from the consortium's studies publicly available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen centers enrolled 83 participants and randomized 82 participants(one participant voluntarily withdrew prior to randomization) who had experienced clinically isolated syndrome and were at risk for developing Multiple Sclerosis (MS) (two or more lesions on Magnetic Resonance Image (MRI) scans) between February 14, 2005 and July 24, 2007.
Pre-assignment Details: At a screening visit, participants underwent procedures to establish that all inclusion criteria were met and none of the exclusion criteria were met. Participants then signed an informed consent form.
Groups:
- Atorvastatin: Drug: Atorvastatin
- Placebo: Non-Active Comparator
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 50 (Safety Sample: 49; Intent-to-Treat Sample: 49; Per Protocol Sample: 39) | 32 (Safety Sample: 32; Intent-to-Treat Sample: 32; Per Protocol Sample: 28)
Completed | 36 | 25
Not Completed | 14 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Primary endpoint met. | 1 | 0
Not completed — Started other MS therapy due to disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 50 | 32 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.4) | 33.9 (8.6) | 33.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 23 | 63
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 46 | 29 | 75
  Canada | 4 | 3 | 7
Number of T2 Lesions at Baseline [Mean (Standard Deviation); unit: Lesion Count] — Number of T2 lesions[1] at baseline. A higher score indicates more severe disease.
  [1] A T2 lesion is defined as an abnormal, hyperintense white-matter area visible on T2 weighted images. Each T2 lesion is visible on at least one brain slice with a surface area ≥ 3mm^2 in plane
  Lesion Count | 21.6 (17.6) | 19.5 (16.5) | 20.8 (17.1)
Number of Gd+ Lesions at Baseline [Mean (Standard Deviation); unit: Lesion Count] — Number of gadolinium-enhancing (Gd+)[1] lesions at baseline. A higher score indicates more severe disease.
  [1]Gd+ lesions are measured on T1 weighted images after injection of 0.1 mM/kg of gadolinium pentate.
  Lesion Count | 0.7 (2.7) | 0.2 (0.5) | 0.5 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of ≥ 3 New T2 Lesions With or Without Gd+ Enhancement or Clinical Exacerbation Through 12 Months.
Description: The occurrence of ≥ T2 lesions[1] with or without gadolinium lesion (Gd+) enhancement[2] or clinical exacerbation[3] through 12 months. A higher score indicates more severe disease
  1. A new T2 lesion is an abnormal, hyperintense white-matter area visible on T2 weighted images that were not present on the baseline scan
  2. A Gd+ enhancement is defined as a contrast enhancement visible on a new T2 lesion
  3. A clinical exacerbation is a new neurological symptom that lasts more than 48 hours in a participant who has been neurologically stable for 30 days following start of study medication
Time Frame: 12 months post-randomization
Population: Intent-to-Treat
Measure: Number; unit: Participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 49 | 32
Participants | 26 | 18
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; This is the primary analysis of the primary endpoint; Test type: Superiority or Other; p = 0.929, Log Rank
Statistical Analysis 2: Comparison: Atorvastatin vs Placebo; This is the secondary analysis of the primary endpoint; Test type: Superiority or Other; p = 0.823, Fisher Exact

2. Secondary Outcome: Proportion of Participants Who Are Diagnosed With Multiple Sclerosis According to the McDonald Criteria
Description: Number of participants diagnosed with Multiple Sclerosis (MS) according to the McDonald criteria[1]
  1. The McDonald criteria uses dissemination in time and space[2] established by Magnetic Resonance Image (MRI) findings to provide a clinical diagnosis for MS
  2. Dissemination in time is established by a new T2 or gadolinium-enhancing (Gd+) lesion found on a repeat MRI. The presence of any 3 of the following establishes dissemination in space: 1 Gd+ lesion or 9 T2 bright lesions if there is no enhancement; ≥1 infratentorial lesion; ≥1 juxtacortical lesion; ≥3 periventricular lesions
Time Frame: 12 months post-randomization
Population: Intent-to-Treat
Measure: Number; unit: Participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 49 | 32
Participants | 29 | 24
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p = .208, Log Rank

3. Secondary Outcome: Proportion of Participants Diagnosed With Multiple Sclerosis According to the McDonald Criteria
Description: as for outcome 2
Time Frame: 18 months post-randomization
Population: Intent-to-Treat
Measure: Number; unit: Participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 49 | 32
Participants | 37 | 24
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority or Other; p = 0.526, Log Rank

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Atorvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/51 | 1/32
Other Adverse Events (participants affected / at risk) | 48/51 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=51) | Placebo (N=32)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=51) | Placebo (N=32)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 1 (2)
Eye pain (Eye disorders) | 2 (6) | 4 (5)
Vision blurred (Eye disorders) | 6 (9) | 5 (9)
Nausea (Gastrointestinal disorders) | 14 (14) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Asthenia (General disorders) | 9 (10) | 5 (6)
Disease progression (General disorders) | 23 (27) | 19 (22)
Fatigue (General disorders) | 14 (16) | 8 (9)
Influenza like illness (General disorders) | 7 (9) | 9 (14)
Bronchitis (Infections and infestations) | 2 (2) | 3 (4)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (5)
Sinusitis (Infections and infestations) | 4 (5) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 8 (16) | 8 (11)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (7)
Alanine aminotransferase increased (Investigations) | 9 (18) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (14) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (3)
C-reactive protein increased (Investigations) | 3 (3) | 2 (2)
Low density lipoprotein decreased (Investigations) | 13 (18) | 1 (1)
Low density lipoprotein increased (Investigations) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (9)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11) | 4 (6)
Dizziness (Nervous system disorders) | 7 (8) | 5 (6)
Headache (Nervous system disorders) | 12 (17) | 7 (10)
Hypoaesthesia (Nervous system disorders) | 20 (41) | 16 (26)
Migraine (Nervous system disorders) | 5 (5) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 3 (4) | 3 (3)
Paraesthesia (Nervous system disorders) | 13 (15) | 8 (14)
Anxiety (Psychiatric disorders) | 5 (6) | 1 (1)
Depression (Psychiatric disorders) | 8 (8) | 10 (10)
Insomnia (Psychiatric disorders) | 11 (11) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No